CLINICAL TRIAL: NCT01811459
Title: Randomized Controlled Trial Comparing Haloperidol, Quetiapine and Placebo in the Pharmacological Treatment of Delirium : The Haloquet Trial
Brief Title: Trial Comparing Haloperidol, Quetiapine and Placebo in the Pharmacological Treatment of Delirium
Acronym: Haloquet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Quebec Firefighters Foundation for Burns (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE12.189
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2016-07

CONDITIONS: Delirium
Keywords: Delirium; ICU; Burn patients; Antipsychotics; Haloperidol; Quetiapine
MeSH Terms: conditions — Delirium | interventions — Quetiapine Fumarate; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Quetiapine (Experimental): Drug: Quetiapine 50-250 mg PO BID (5 levels of treatment) + IV Placebo Rescue IV haloperidol available.
  Interventions: Drug: Quetiapine
- Haloperidol (Experimental): Drug: Haloperidol 1-5 mg BID (5 levels of treatment) + PO placebo Rescue IV haloperidol available.
  Interventions: Drug: Haloperidol
- Placebo (Placebo Comparator): IV placebo + PO placebo Rescue IV haloperidol available.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine — PO
  Arms: Quetiapine
Drug: Haloperidol — IV
  Arms: Haloperidol
Drug: Placebo — PO or IV
  Arms: Placebo

SUMMARY:
Background:

Delirium is an important problem in critical care. Its prevalence often reaches 75% in intensive care patients. Its occurrence is associated with numerous complications and deleterious consequences such as death, longer stay, higher cost, and long-term cognitive impairment. Delirium treatment entails correcting its underlying causes and usually initiating a pharmacological intervention with an antipsychotic. Typical antipsychotics, particularly haloperidol, are commonly used to treat delirium although few placebo-controlled trials of pharmacological treatments for delirium have been conducted. Furthermore, appropriate doses for delirium treatment have yet to be established. In critical care, two pilot studies provided the first randomized, placebo-controlled evidence for the pharmacologic treatment of ICU delirium. One found that neither haloperidol nor ziprasidone significantly reduced the incidence or duration of delirium compared with placebo whereas the other one found that quetiapine added to as-needed haloperidol resulted in faster delirium resolution.

Objective:

The goal of this study is to determine the effectiveness of antipsychotics in regular dosage regimen (quetiapine group and haloperidol group) compared to as-needed haloperidol (placebo group) in the pharmacological treatment of delirium. We will conduct a three-arm randomized controlled trial to achieve this goal.

Materials and Methods:

During one year, 45 delirious patients from three intensive care units will be recruited and randomized into one of three groups. Randomization will be performed in blocks of 9 by the pharmacy department, using a random numbers table.

Patients will be continuously screened for delirium using the Intensive Care Delirium Screening Checklist (ICDSC) as part of routine care. A positive screening score (≥4) will warrant confirmation of delirium diagnosis by the treating physician. Treatment will begin according to randomization group, provided that informed consent has been obtained. Delirium status will be monitored during the episode using the Nursing Delirium Screening Scale (Nu-DESC). When the Nu-DESC monitoring will become negative for delirium (total score below 2), the resolution of the episode will be confirmed by the treating physician. A clinical evaluation by a psychiatrist will be performed within 24-48 hours of each of the two evaluations made by the treating physician (beginning and end of the delirium episode).

The treating physician will initiate twice-daily treatment at the first of five levels for each of the three groups: 1) 1 mg of intravenous (IV) haloperidol + oral (PO) placebo, 2) 50 mg of PO quetiapine + IV placebo, or 3) IV + PO placebo. Therapy will be titrated upwards on a daily basis by increments of 1) 1 mg of IV haloperidol or 2) 50 mg of PO quetiapine, or 3) IV + PO placebo every 12 hrs, respectively, if the subject received at least two doses of as-needed haloperidol in the previous 24 hrs. As-needed (PRN) doses of 2 mg of IV haloperidol q 30 minutes will be available to patients from all three groups and administered by nurses until symptoms associated with delirium resolve. In case of unsuccessful as-needed treatment, rescue (STAT) doses of 5 mg of IV haloperidol q 30 minutes will be available to patients from all three groups and will be administered by nurses if agreement is reached with the treating physician that the situation indeed calls for it. The treatment level of patients requiring a STAT dose will immediately be raised to the above level. The treatment will stop when one of the following occurs: (1) the subject is deemed by the treating physicians, based on their clinical judgment, to no longer demonstrate signs of delirium and, therefore, to no longer require scheduled therapy with an antipsychotic agent; (2) 21 days of therapy has elapsed; (3) ICU discharge occurred; or (4) a life-threatening adverse event potentially attributable to the study drug occurred that warranted discontinuation of the study drug.

Adverse effects will be closely monitored: extrapyramidal reactions, neuroleptic malignant syndrome, drowsiness, hypotension, QTc prolongation. The treatment level of patients presenting a non life-threatening adverse event will immediately be lowered to the level directly below.

The sample size was calculated for a 2-tailed test with an alpha of .05 and a power of .80.

The primary statistical analysis will involve Cox proportional time to event analysis comparing the three groups. Secondary analysis will use T-test comparisons for continuous variables and chi square for proportional analysis.

DETAILED DESCRIPTION:
Primary Outcome Measures:

•Time to first resolution of delirium.

Secondary Outcome Measures:

* Days in delirium during the study
* Duration of delirium
* Severity of delirium (highest Nu-DESC score, mean episode Nu-DESC score)
* ICU and hospital mortality
* ICU and hospital length of stay
* Length of mechanical ventilation
* Time spent deeply sedated (RASS <3)
* Episodes of subject-initiated device removal
* Use of haloperidol therapy (including total dose in haloperidol equivalents during the study, number of doses, number of days of therapy, use of rescue IV haloperidol)
* Average daily and maximum total antipsychotic drug dose in haloperidol equivalents
* Duration of study drug administration
* Use of benzodiazepines (converted to lorazepam equivalents)
* Use of opioids (converted to morphine equivalents)
* QTc prolongation
* Extrapyramidal symptoms
* Neuroleptic malignant syndrome

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients with a diagnosis of delirium made by a psychiatrist.

Exclusion Criteria:

* Patients with active schizophrenia or bipolar disorder.
* Patients with Parkinson disease.
* Patients with severe liver failure.
* Patients with alcohol or sedative/hypnotics dependence.
* Patients with QTc interval above 500 msec.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Time to first resolution of delirium | 21 days
  Confirmed by clinical evaluation of a psychiatrist

SECONDARY OUTCOMES:
Days in delirium during the study | 21 days
  From log
Duration of delirium | 21 days
  From log
Severity of delirium (highest Nu-DESC score, mean episode Nu-DESC score) | 21 days
  Nursing evaluation every 8 hours- shift
ICU and hospital mortality | 21 days
  From the chart
ICU and hospital length of stay | 21 days
  From the chart
Length of mechanical ventilation | 21 days
  From daily clinical évaluation
Time spent deeply sedated (RASS <3) | 21 days
  From chart
Episodes of subject-initiated device removal | 21 days
  From daily clinical évaluation
Use of haloperidol therapy (including total dose in haloperidol equivalents during the study, number of doses, number of days of therapy, use of rescue IV haloperidol) | 21 days
  From long
Average daily and maximum total antipsychotic drug dose in haloperidol equivalents | 21 days
  From long
Duration of study drug administration | 21 days
  From log
Use of benzodiazepines | 21 days
  All benzodiazepines received in lorazepam equivalent
Use of opioids | 21 days
  All opioids received in morphine équivalent
QTc prolongation | 21 days
  From EKG recording
Extrapyramidal symptoms | 21 days
  Daily clinical evaluation
Neuroleptic malignant syndrome | 21 days
  Daily clinical evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes